CLINICAL TRIAL: NCT05478369
Title: The Effect of Reading Story Books on Children's Preoperative Fear and Anxiety Levels
Brief Title: The Effect of Reading Story Books on Fear and Anxiety Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ARZU SARIALİOĞLU, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/554
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Operative Incision
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- storybook (Experimental): anxiety and fear
  Interventions: Behavioral: storybook
- control (No Intervention): not anxiety and fear

INTERVENTIONS:
Behavioral: storybook — anxiety and fear during operative
  Arms: storybook

SUMMARY:
The aim of this project is to determine the effect of reading the story book, which is considered within the scope of the pedagogically approved research that introduces the surgical environment before the surgical intervention in children, on the pain and anxiety of the child. The project is a randomized controlled trial. The population of the research will be children between the ages of 4 and 6 who come to Atatürk University Health Research and Application Center Pediatric Surgery Clinic between March and September 2022 for treatment. The research sample; children and parents who are hospitalized in the clinic on the dates specified by the probabilistic sampling method and meet the research criteria, willing to participate in the research. "Survey Form", "Modified Yale Preoperative Anxiety Scale (mYPAS)" and "Child Fear Scale" will be used in data collection.

DETAILED DESCRIPTION:
Type of Study: The study is of the randomized controlled experimental type. Place and Time of the Research: The research will be carried out between March-September 2022 at Atatürk University Health Research and Application Center Pediatric Surgery Clinic. Surgical procedures performed in the clinic are frequently prepuce, hernias, undescended testis, acute abdominal traumas and dilatation.

Population and Sample of the Study: The population of the research will be children aged 4-6 years who come to Atatürk University Health Research and Application Hospital Pediatric Surgery Clinic between March-September 2022 for treatment.

The research sample; hernia and undescended testis will be operated on the dates specified by the probabilistic sampling method and children who meet the research criteria and volunteer to participate in the research will be formed.

In order to prevent interaction between the groups of children in the clinic, data collection will not be carried out simultaneously in the story group and control groups. In order to ensure randomization, children who met the criteria will be included in the control group in the first week, and children who come in the second week will be included in the story group, and this cycle will be continued until the end of the study and randomization will be ensured.

Data Collection Tools: Questionnaire Form, Modified Yale Preoperative Anxiety Scale and Child Fear Scale will be used to collect research data. The book titled "Elif Is Surgery", which is licensed by Çamlıca Children's Publishing, which owns the copyrights, will be used as an intervention tool in the research.

Questionnaire Form: In this form, which was prepared by the researcher by examining the literature; There will be questions about the introductory features of the child and the parent.

Modified Yale Preoperative Anxiety Scale (mYPAS): The Yale Preoperative Anxiety Scale (YPAS), which was developed in 1995 to measure the preoperative anxiety of children, was modified in 1997 (mYPAS) and used in many studies covering various health fields such as dentistry, anesthesia, surgery, and pediatrics. The scale evaluates five basic parameters. These; Activity includes speech, emotional state, marked arousal, and relationship with family. In the scale, the parameters of activity, emotional state, marked arousal state and relationship with family are evaluated between (1-4) and speech (1-6).

Child Fear Scale (CFS): Child Fear Scale was developed in 2011 to measure fear in children undergoing painful medical procedures. The Child Fear Scale is a scale from 0-4 showing five faces ranging from a neutral expression (0 = no worry) to the feared face (4 = serious anxiety).

Intervention Tool to be Used in Research Storybook: As an intervention tool in the research, the book titled "Elif Is Surgery" will be read by her parents.

In the selection of the story book, attention was paid to the fact that it was pedagogically appropriate and at the same time the author of the book was a child developmentalist and pedagogue. In this storybook, the operating environment is introduced in a way that children can understand and is suitable for the age group of the study. Words such as cut and blood, which are specific to this age, are not used in the storybook. While the story book will be read, the child's opinion will be taken and the book will be read with a character name that he wants. For example, ask the children, "What name would you like to give your character before the book is read?" Asking the child's opinion will increase his self-confidence, and at the same time, it will be ensured that he listens carefully to the story with the curiosity of "What will happen to my character?" Data Collection The researcher will be in the pediatric surgery service for 2 days to examine the pediatric surgery service and will make a preliminary application before collecting the data of the children in the storybook group and the control group children. The children and their parents were given preliminary information about the research (the purpose of the research, why the research was conducted, the story book would be used to relieve the child's fear and anxiety, it was thought that it would be effective in preventing fear, etc.) will be obtained through face-to-face interviews.

Control Group: Questionnaires and scales will be filled by the researcher 30 minutes before the surgery. Only routine applications will be done within 5 minutes. The scales will be refilled 10 minutes before the surgery and when the child moves to the premedication room. The families of the children will be with the children until the premedication room. Filling out the forms will take 5-10 minutes on average.

Story Group: Questionnaires and scales will be filled in 30 minutes before the surgery by the researcher. The child's parent will read the storybook. In reading the story book; It will reduce fear and anxiety by attracting the patient's attention (sound, image…) and enabling him to get away from the negative emotions he is in. Routine applications will be done within 5 minutes. The scales will be refilled 10 minutes before the surgery and when the child moves to the premedication room. The families of the children will be with the children until the premedication room. Filling out the forms will take 5-10 minutes on average.

Evaluation of Data The processing and statistical analysis of the collected data will be done with the analysis software called SPSS (Statistical Package for the Social Sciences) for Windows 20.0.

Ethical Principles of Research In order to carry out the research, official permission from the relevant institution will be obtained from the Ethics Committee with ethical approval. Children who meet the criteria of the research group will be informed about the purpose of the study, their questions will be answered, and their verbal and written consent will be obtained. Parents and children will be informed that the data collected during the research will be processed anonymously, confidentially, and will not be used outside of the study in question, and that they can leave the study whenever they wish. Since the research is based on the use of data obtained from humans, and therefore, due to the necessity of observing personal rights, the relevant ethical principles "Informed Consent", "Volunteerism" and "Protection of Confidentiality" will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 4-6
* Hernias, undescended testis surgery
* Does not have a disability related to developmental areas
* parent's literacy

Exclusion Criteria:

* Not between 4-6 years old
* No hernias, undescended testis surgery
* Having a disability related to developmental areas
* parent's illiteracy

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2022-03-19 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Child Fear Scale (CFS) | 9 MONTHS
  The scale was developed in 2011. The Child Fear Scale is used to determine the level of fear in children undergoing painful medical procedures. The Child Fear Scale is a scale from 0-4 showing five faces ranging from a neutral expression (0 = no worry) to the feared face (4 = serious anxiety).
Modified Yale Preoperative Anxiety Scale (mYPAS) | 9 MONTHS
  Yale Preoperative Anxiety Scale (YPAS), which was developed in 1995 to measure children's preoperative anxiety, was modified in 1997 (mYPAS) and used in many studies covering various health fields such as dentistry, anesthesia, surgery, and pediatrics. The scale evaluates five basic parameters. These; Activity includes speech, emotional state, marked arousal, and relationship with family. In the scale, the parameters of activity, emotional state, marked arousal state, and family relationship are evaluated between (1-4) and speech (1-6).

CONTACTS AND LOCATIONS:
Overall Officials: ARZU SARIALİOĞLU, PHD, Study Director — Ataturk University
Locations (1):
- Ataturk University Nursing of Faculty, Erzurum, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
THE ARTICLE IS INTENDED TO BE SHARED AFTER IT IS PUBLISHED

REFERENCES:
- [Derived] Sarialioglu A, Kurudirek F, Oluc T. The effect of storybook reading on children's preoperative fear and anxiety levels: A randomized controlled study. Child Care Health Dev. 2023 Sep;49(5):906-913. doi: 10.1111/cch.13100. Epub 2023 Feb 8. PMID 36735635